CLINICAL TRIAL: NCT05528029
Title: International Ledless Pacemaker Registry (i-LEAPER)
Brief Title: International Ledless Pacemaker Registry
Acronym: i-LEAPER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Luigi Sacco University Hospital (Other)
Collaborators: Università degli Studi di Brescia (Other); Centro Cardiologico Monzino (Other); University Hospital, Zürich (Other); Azienda Ospedaliera Cardinale G. Panico (Other); Azienda Ospedaliera San Gerardo di Monza (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); San Raffaele University Hospital, Italy (Other); Ospedale V. Fazzi (Other); Ospedali Riuniti Ancona (Other); Universitair Ziekenhuis Brussel (Other); Università degli Studi di Ferrara (Other); University of Padova (Other)
Responsible Party: Principal Investigator, Giovanni B Forleo, Section Head Electrophysiology and Clinical Pacing, Luigi Sacco University Hospital
Other Study IDs: Hsacco2022
Record Dates: First submitted 2022-08-31; First posted 2022-09-06 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Block Complete Heart; Atrial Fibrillation
Keywords: leadless pacing
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Leadless Pacemaker (Micra) — Micra leadless pacemaker is implanted in the right ventricle via femoral vein. The Micra introducer/dilator assembled system is inserted over a stiff guidewire in the right atrium. After the removal of the guidewire and the dilator, the delivery system is advanced into the introducer and the Micra is placed under fluoroscopy guidance, preferably in the septal region of the right ventricle.

SUMMARY:
The Micra MC1VR01 or Micra AVMC1AVR1 Transcatheter Pacing System (Medtronic, Inc., Minneapolis, MN, USA) has become a major breakthrough as an alternative to standard transvenous pacemakers.

The aim of this multi-center study is to assess the clinical outcomes of patients implanted with Micra LLPM in real life, in different clinical scenarios.

DETAILED DESCRIPTION:
The study includes consecutive patients implanted with a pacemaker leadless device (Micra Transcatheter Pacing System; Medtronic, Inc., Minneapolis, MN, USA).

Baselines characteristics, procedural and clinical outcomes will be collected and analyzed.

ELIGIBILITY:
Inclusion Criteria: All patients implanted with the MIcra leadless pacing system

* At least 1 month of follow up
* At least 1 post-implantation assessment, in accordance to the routine clinical practice of every center

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in whom a MIcra was implanted for a cardiac bradyarrhythmia.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause mortality | through study completion, an average of 2 years
  overall mortality
Implant complication rates | during and immediately after the intervention
  Dislodgments, Cardiac perforation, vascular complications (access site).
Electrical performance of the pacing system | Through study completion, an average of 2 years
  Pacing thresholds
Electrical performance of the pacing system | Through study completion, an average of 2 years
  R wave sensing
Electrical performance of the pacing system | Through study completion, an average of 2 years
  pacing impedances values
Upgrading with a different pacing system | Through study completion, an average of 2 years
  Need of an additional transvenous pacing system

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni B Forleo, MD, PhD, Principal Investigator — Luigi Sacco University Hospital; Gianfranco MItacchione, MD, PhD, Principal Investigator — Luigi Sacco University Hospital
Locations (12):
- Heart Rhythm Management Centre, Universitair Ziekenhuis Brussel, Postgraduate program in Cardiac Electrophysiology and Pacing, European Reference Networks Guard-Heart, Vrije Universiteit, Brussels, Belgium
- Italy (10):
  - Cardiology and Arrhythmology Clinic, University Hospital "Umberto I-Salesi-Lancisi", Ancona (IT), Ancona
  - Department of Cardiology, IRCCS, Azienda Ospedaliero Universitaria Di Bologna, Policlinico Di S. Orsola, Bologna
  - Spedali Civili di Brescia, Brescia
  - Cardiology Unit, Vito Fazzi Hospital, Lecce (IT), Lecce
  - Arrhythmology and Electrophysiology Unit, San Raffaele Hospital, IRCCS, Milan
  - Azienda Ospedaliera - Polo Universitario - "Luigi Sacco", Milan
  - Department of Clinical Electrophysiology and Cardiac Pacing, Centro Cardiologico Monzino, IRCSS, Milan
  - Department of Cardiology, ASST Monza, San Gerardo Hospital, Monza
  - Departtment of Cardiac, Thoracic Vascular Sciences and Public Health University of Padova, Padua
  - Cardiology Unit, "Card. G. Panico" Hospital, Tricase (IT), Tricase
- University Hospital Zurich,, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Reynolds D, Duray GZ, Omar R, Soejima K, Neuzil P, Zhang S, Narasimhan C, Steinwender C, Brugada J, Lloyd M, Roberts PR, Sagi V, Hummel J, Bongiorni MG, Knops RE, Ellis CR, Gornick CC, Bernabei MA, Laager V, Stromberg K, Williams ER, Hudnall JH, Ritter P; Micra Transcatheter Pacing Study Group. A Leadless Intracardiac Transcatheter Pacing System. N Engl J Med. 2016 Feb 11;374(6):533-41. doi: 10.1056/NEJMoa1511643. Epub 2015 Nov 9. PMID 26551877
- [Derived] Mitacchione G, Schiavone M, Gasperetti A, Arabia G, Breitenstein A, Cerini M, Palmisano P, Montemerlo E, Ziacchi M, Gulletta S, Salghetti F, Russo G, Monaco C, Mazzone P, Hofer D, Tundo F, Rovaris G, Russo AD, Biffi M, Pisano ECL, Chierchia GB, Della Bella P, de Asmundis C, Saguner AM, Tondo C, Forleo GB, Curnis A. Outcomes of leadless pacemaker implantation following transvenous lead extraction in high-volume referral centers: Real-world data from a large international registry. Heart Rhythm. 2023 Mar;20(3):395-404. doi: 10.1016/j.hrthm.2022.12.002. Epub 2022 Dec 7. PMID 36496135